CLINICAL TRIAL: NCT02802176
Title: Randomized Controlled Trial Comparing Intra-vaginal Culture of Embryos Using INVOcell Device to In-vitro Culture of Embryos Using Minimal Stimulation Protocols
Brief Title: Comparing Intra-vaginal Culture of Embryos to In-vitro Culture of Embryos With Minimal Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment and completion of screening qualifiers.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 166094
Record Dates: First submitted 2016-06-12; First posted 2016-06-16 (Estimated); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Arm 1: intra-vaginal culture using INVOcell device. Arm 2: Traditional In-Vitro Fertilization (IVF) culture in an embryology laboratory
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intra-vaginal culture - INVOcell device (Experimental): 3 day intra-vaginal incubation using the INVOcell device
  Interventions: Device: INVOcell device
- Traditional IVF culture (Active Comparator): 3 day traditional IVF incubation
  Interventions: Other: Traditional IVF

INTERVENTIONS:
Device: INVOcell device — intra-vaginal culture of embryos using INVOcell device
  Arms: Intra-vaginal culture - INVOcell device
Other: Traditional IVF — traditional culture of embryos in-vitro
  Arms: Traditional IVF culture

SUMMARY:
The purpose of this study is to evaluate implantation rate with intra-vaginal culture (IVC) with the INVOcell device versus traditional In-Vitro Fertilization (IVF) while using minimal stimulation protocols

DETAILED DESCRIPTION:
This is a Phase IV, single center randomized controlled trial evaluating intra-vaginal culture (IVC) using INVOcell versus traditional In-Vitro Fertilization (IVF) using oral stimulation or minimal gonadotropin stimulation protocols. The pilot aims to includes 40 women who will be randomized to either the intra-vaginal culture group (N=20) using INVOcell or to the traditional IVF group (N=20).

Primary aim is implantation rate, which is defined by number gestational sacs seen on early pregnancy ultrasound divided by number of embryos transferred.

Secondary aims are:

* Embryo quality, which is measured by system similar to the Gardner grading system at cleavage stage. Reported quality will be converted to the simplified SART embryo scoring system which provides an overall categorical embryo grade of "Good", "Fair" or "Poor".
* Fertilization rate, which is defined by the total number of fertilized oocytes divided by total number of mature oocytes retrieved. This comparison will take place on day-3, as that is when the IVC embryos will be assessed.
* Clinical pregnancy rate, which is defined by the number of fetal poles with heartbeat seen on ultrasound divided by the number of embryos transferred.
* Live birth rate, which is defined by the number of living babies delivered divided by the number of transfers

ELIGIBILITY:
Inclusion Criteria:

* Normal uterine cavity
* One or more years of infertility
* Normal male partner semen analysis

Exclusion Criteria:

* Age <18 years old or >37 years old
* Antral Follicle Count (AFC) <8
* Abnormal male partner semen analysis or use of donor sperm
* Vaginal inflammation or genital (vaginal, uterine, tubal) infection
* Uncontrolled chronic disease (such as uncontrolled diabetes or hypertension)
* Uterine anatomic abnormalities
* Allergy to plastics or inability to use diaphragm retention device
* Untreated hydrosalpinx
* Current alcohol abuse (defined by >14 drinks/week)
* Prior history of IVF cycle where fertilization did not occur
* History of recurrent pregnancy loss

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelle Cedars, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco - Center for Reproductive Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: INVOcell device — http://www.invobioscience.com/
- See also: University of California San Francisco Center for Reproductive Health — https://crh.ucsf.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between October 2016 to February 2022, apart from a two year period of the COVID-19 Pandemic. Potential subjects were recruited from patient populations of the UCSF Center for Reproductive Health, the Zuckerberg San Francisco General Hospital and the general public.
Pre-assignment Details: 9 of 39 enrolled participants screen failed out of the study prior to randomization assignment. 6 never moved forward with starting clinical fertility treatment, 1 responded poorly to the minimal stimulation medication protocol that was part of the study design and couldn't proceed with the egg retrieval procedure, 1 was at risk for mild Ovarian Hyperstimulatory Syndrome and 1 voluntarily dropped out of the study prior to randomization due to financial and insurance coverage reasons.
Period: Overall Study
Arm/Group | Traditional IVF Culture | Intra-vaginal Culture - INVOcell Device
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Intra-vaginal Culture - INVOcell Device: 3 day intra-vaginal incubation of embryos using INVOcell device
- Active Comparator: Traditional IVF Culture: 3 day traditional In Vitro Fertilization embryo incubation
- Total: Total of all reporting groups
Arm/Group | Experimental: Intra-vaginal Culture - INVOcell Device | Active Comparator: Traditional IVF Culture | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Implantation Rate
Description: defined by number gestational sacs seen on early pregnancy ultrasound typically done at 6 weeks of gestational age divided by number of embryos transferred
Time Frame: approximately 4 weeks following randomization. Clinically this is typically done around 6 weeks of gestational age
Population: 3 participants in the Traditional IVF culture arm and 2 participants in the intra-vaginal culture arm were excluded from analysis as they did not undergo embryo transfers.
Measure: Mean (Standard Deviation); unit: percentage of embryo transfers
Arm/Group | Intra-vaginal Culture - INVOcell Device | Traditional IVF Culture
Number analyzed (Participants) | 12 | 13
percentage of embryo transfers | 12.50 (0.2976) | 42.31 (43.17)

2. Secondary Outcome: Embryo Quality
Description: -Embryo quality, which is measured by system similar to the Gardner grading system at cleavage stage. Reported quality will be converted to the simplified SART embryo scoring system which provides an overall categorical embryo grade of "Good", "Fair" or "Poor".
Time Frame: measured after 3 days of incubation
Population: 1 participant from the intra-vaginal culture arm and 2 participants from the traditional IVF culture arm were excluded from the analysis due fertilization failures and no embryos on culture day 3 to grade.
Measure: Count of Units; unit: Culture day 3 cleavage-stage embryos
Units Other Than Participants: Culture day 3 cleavage-stage embryos
Arm/Group | Intra-vaginal Culture - INVOcell Device | Traditional IVF Culture
Number analyzed (Participants) | 13 | 14
Number analyzed (Culture day 3 cleavage-stage embryos) | 45 | 58
Culture day 3 cleavage-stage embryos
  "Good" | 34 | 48
  "Fair" | 4 | 4
  "Poor" | 7 | 6

3. Secondary Outcome: Fertilization Rate
Description: defined by the total number of fertilized oocytes divided by total number of mature oocytes retrieved
Time Frame: measured after 3 days of incubation
Measure: Mean (Standard Deviation); unit: percentage of oocytes fertilized
Arm/Group | Intra-vaginal Culture - INVOcell Device | Traditional IVF Culture
Number analyzed (Participants) | 14 | 16
percentage of oocytes fertilized | 61.75 (25.19) | 63.4 (30.55)

4. Secondary Outcome: Clinical Pregnancy Rate
Description: which is defined by the number of fetal poles with heartbeat seen on early pregnancy ultrasound typically done at 6 weeks of gestational age divided by the number of embryos transferred
Time Frame: approximately 4 weeks following randomization. Clinically this is typically done around 6 weeks of gestational age
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of embryo transfers
Arm/Group | Intra-vaginal Culture - INVOcell Device | Traditional IVF Culture
Number analyzed (Participants) | 12 | 13
percentage of embryo transfers | 12.5 (29.76) | 46.15 (45.83)

5. Secondary Outcome: Live Birth Rate
Description: which is defined by the number of living babies delivered divided by the number of transfers
Time Frame: 9 months after embryo transfer
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of embryo transfers
Arm/Group | Intra-vaginal Culture - INVOcell Device | Traditional IVF Culture
Number analyzed (Participants) | 12 | 13
percentage of embryo transfers | 12.5 (29.76) | 38.46 (44.52)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Intra-vaginal Culture - INVOcell Device | Traditional IVF Culture
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

LIMITATIONS AND CAVEATS:
Due to capacity limitations of the INVOcell device, participants in each arm were only allowed to fertilize up to 7 oocytes. Excess oocytes were frozen for all subjects for future use. This study also used a mild stimulation medication protocol to limit excessive eggs being produced under the assumption few participants would reach this imposed limit. At the time of study design, the device was only FDA approved for up to 3 day of embryo culturing. These factors may have limited some findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02802176/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT02802176/ICF_001.pdf